CLINICAL TRIAL: NCT02056340
Title: Statin Therapy in Acute Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Maureen Chase MD MPH, Principal Investigator, Maureen Chase MD MPH, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P000026; 1K23GM101463-01A1 (NIH); FWA00003245 (Other: BIDMC)
Record Dates: First submitted 2013-10-15; First posted 2014-02-06 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): Patients will be administered study medication (atorvastatin 40 mg) orally once daily for 5 days, for a maximum of 7 days for those who remain hospitalized.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Patients will be administered study medication (matched placebo) orally once daily for 5 days, for a maximum of 7 days for those who remain hospitalized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Influenza (the 'flu') is a common virus infecting approximately 5-20% of the population in the United States and causing as many as 500,000 deaths worldwide each year. Currently, there are only a few treatments for influenza infection and none of these target inflammation that can be caused by the virus. This study will test whether the anti-inflammatory effects of statins, a class of drugs most often used to treat high cholesterol, will decrease the severity of illness in patients who are infected with influenza by testing markers of inflammation in the blood and recording resolution of influenza illness.

ELIGIBILITY:
Inclusion Criteria:(all must be present):

1. Adult patient (age > 18 years)
2. Positive influenza DFA/RAT test result
3. <12 hours from positive influenza test result

Exclusion Criteria:

1. Prior statin medication use (within 30 days of positive influenza test result)
2. Comfort measures only designation or anticipated withdrawal of life-support
3. Atorvastatin specific exclusions:

   1. Documented liver cirrhosis or liver dysfunction (AST or ALT greater than 240)
   2. Known allergy or intolerance to statins
   3. Rhabdomyolysis (CPK elevation > 6x normal)
   4. Patients taking the following medications: cyclosporine, HIV protease inhibitors, hepatitis C protease inhibitor telaprevir, fibric acid derivatives (gemfibrozil), niacin, azole antifungals (itraconazole, ketoconazole) clarithromycin and colchicine
4. Patients unable to take oral or nasogastric medications or plan for no oral intake as part of medical course (eg. emergent surgical intervention)
5. Known pregnancy or active breastfeeding
6. Inability to provide written informed consent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Chase, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- The Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chase M, Cocchi MN, Grossestreuer AV, Liu X, Vine J, Moskowitz AL, Donnino MW. Randomized Controlled Trial of Atorvastatin in Acute Influenza in the Emergency Department. West J Emerg Med. 2025 Apr 29;26(3):600-608. doi: 10.5811/westjem.33580. PMID 40561994

RESULTS

PARTICIPANT FLOW:
Groups:
- Atorvastatin: Patients will be administered study medication (atorvastatin 40 mg) orally once daily for 5 days, for a maximum of 7 days for those who remain hospitalized.
  Atorvastatin
- Placebo: Patients will be administered study medication (matched placebo) orally once daily for 5 days, for a maximum of 7 days for those who remain hospitalized.
  Placebo
Period: Overall Study
Arm/Group | Atorvastatin | Placebo
Started | 59 | 57
Completed | 52 | 46
Not Completed | 7 | 11
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin | Placebo | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [23 to 51] | 43 [29 to 58] | 37 [25 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 39 | 72
  Male | 26 | 18 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 40 | 74
  Black/ African American | 20 | 15 | 35
  Other | 4 | 2 | 6
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.2 [23.4 to 33.9] | 28.4 [26.4 to 33.4] | 28.1 [23.8 to 33.5]

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Markers From Time Zero to 72 Hours
Description: The primary IL- 6 measurements were at time zero and at 72 hours. Analysis was performed using a linear mixed effects model to make use of all biomarker timepoints as hospitalized patients had biomarkers measured at additional timepoints.
Time Frame: Baseline to 72 hours
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 51 | 48
pg/ml
  Baseline | 2.4 [.072 to 5.27] | 3.46 [1 to 6.84]
  72 hours | 0.91 [0.23 to 2.23] | 0.57 [.031 to 1.58]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; We used a linear mixed-effects model which accounted for all measurements taken and the time that those measurements were taken; Test type: Other; p = 0.611, Mixed Models Analysis — Threshold for significaance was p value <0.05

2. Secondary Outcome: Severity of Illness Score Baseline to 72 Hours
Description: Composite score for 5 major symptoms (fever, cough, sore throat, headache, myalgia) ranked from 0 to 3 (none, mild, moderate, severe) for a score ranging from 0 to 15. Higher scores reflect more severe symptoms.
Time Frame: Baseline and 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Atorvastatin | Placebo
Number analyzed (Participants) | 59 | 57
score on a scale
  Baseline | 8 [6 to 10] | 8 [6 to 11]
  72 hours | 2 [1.5 to 4] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Atorvastatin vs Placebo; The primary comparison was at 72 hours for the self-reported influenza severity score; Test type: Other; p = 0.029, Mixed Models Analysis — P value reflects baseline to 72 hours between groups. A p-value <0.05 will be considered significant

3. Other Pre Specified Outcome: Progression to Shock State
Description: The investigators will assess the effect of statin therapy on rates of development of shock state
Time Frame: From date of randomization until discharge from hospital
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Severity of Illness
Description: The investigators will assess the effect of statin therapy on APACHE II scores
Time Frame: 24 hours post enrollment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: In-hospital Mortality
Description: The investigators will assess the effect of statin therapy on in-hospital mortality
Time Frame: From date of randomization until the date of first documented discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 year
Reporting Status: Not Posted

6. Other Pre Specified Outcome: ICU and Hospital Length of Stay
Description: The investigators will assess the effect of statin therapy on hospital and ICU length of stay.
Time Frame: From date of randomization until the date of ICU discharge (in the event of ICU admission) and/or hospital discharge, based on an estimated average of 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | Atorvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/57
Other Adverse Events (participants affected / at risk) | 4/59 | 5/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin (N=59) | Placebo (N=57)
Safety lab testing AST, ALT and CK levels (Hepatobiliary disorders) | 1 (1) | 2 (2) — CK levels elevated
GI Distress (Gastrointestinal disorders) | 2 (2) | 1 (1) — Patients presenting with GI distress such as gastroenteritis, diarrhea, and yellow stool.
Focal Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Facial tingling (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient complained of worsening nausea and dry heaves.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT02056340/Prot_SAP_000.pdf
  • Informed Consent Form: Part D: Informed Consent (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT02056340/ICF_001.pdf
  • Informed Consent Form: Verbal Consent - Rapid Antigen Test (RAT) (2015-12-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02056340/ICF_002.pdf